CLINICAL TRIAL: NCT01716936
Title: A Retrospective Multicenter Review of Early Onset Spinal Deformity Patients That Underwent Either a Primary or Revision Spinal Bracing Procedure With the Ellipse Technologies MAGEC Spinal Bracing and Distraction System
Brief Title: A Retrospective Review of Early Onset Spinal Deformity Patients Treated With the Ellipse MAGEC System
Status: Completed | Type: Observational
Sponsor: Ellipse Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PR0056
Record Dates: First submitted 2012-09-19; First posted 2012-10-30 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Thoracic Insufficiency Syndrome
Keywords: Thoracic Insufficiency Syndrome; Early Onset Spinal Deformity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MAGEC Implant: All patients implanted with the MAGEC System will be reviewed for inclusion into this retrospective study.

SUMMARY:
The purpose of this study is to determine the safety profile and probable benefit of the Ellipse Technologies Inc. MAGEC System in subjects with early onset spinal deformity associated with thoracic insufficiency syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Early onset spinal deformity with any etiology
* Cobb angle measurement of 30 degrees or greater at the time of primary surgery
* Thoracic spine height (T1 to T12) less than 22 cm at the time of primary surgery
* Age less than 11 years old at the time of MAGEC implant
* Implanted with the MAGEC system as either a primary or secondary revision spinal bracing procedure
* Patient has been implanted for a minimum of 6 months
* Patient signs informed consent for the use of their personal private data

Exclusion Criteria:

* Patient declines to sign informed consent for the use of their personal private data.

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients worldwide implanted with the Ellipse Technologies Spinal Bracing and Distraction System (Invitation to Volunteer Non-Probability Sample).
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in Cobb Angle | Baseline and 6, 12, 18 and 24 Months Postoperatively
  Measured in Degrees
Change in Thoracic Spine Height | Baseline and 6, 12, 18 and 24 Months Postoperatively
  Measured in millimeters (mm)
Change in Space Available for Lung | Baseline and 6, 12, 18 and 24 Months Postoperatively
  Measured as a percentage (%)
Ocurrence of Procedure-Related Complications | Baseline, Device Implant and 6, 12, 18 and 24 Months Postoperatively
Occurrence of Adverse Events | Baseline and 6, 12, 18 and 24 Months Postoperatively

SECONDARY OUTCOMES:
Change in Coronal Balance | Baseline and 6, 12, 18 and 24 Months Postoperatively
  Measured in millimeters (mm)
Change in Sagittal Balance | Baseline and 6, 12, 18 and 24 Months Postoperatively
  Measured in millimeters (mm)
Occurrence of Subsequent surgical interventions following initial implantation | Baseline and 6, 12, 18 and 24 Months Postoperatively
Change in Weight | Baseline and 6, 12, 18 and 24 Months Postoperatively
  Measured in kilograms (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Behrooz A Akbarnia, MD, Principal Investigator — San Diego Center for Spinal Disorders
Locations (15):
- University of Cairo Public Hospital, Cairo, Egypt
- Finland (2):
  - University of Helsinki, Helsinki
  - Turku University Hospital, Turku
- University of Hong Kong, Hong Kong, Hong Kong
- Italy (2):
  - Instituto Rizzoli, Bologna
  - Bambin Gesu, Rome
- Starship Children's Hospital, Auckland, New Zealand
- Turkey (Türkiye) (5):
  - Ankara Gazi Universitesi Hastanesi, Ankara
  - Hacettepe University Hospital, Ankara
  - Florence Nightingale Hospital Ortopedi Bolumu, Istanbul
  - Marmara Üniversitesi Eğt.ve Arş.Hastanesi, Istanbul
  - Ege Sağlık Hastanesi, Izmir
- United Kingdom (3):
  - Royal National Orthopaedic Hospital NHS Trust, Stanmore, Middlesex
  - University Hospital of Wales, Cardiff
  - The Harley Street Clinic, London